CLINICAL TRIAL: NCT03791372
Title: Clinical Effect and Safety of Autologous Umbilical Cord Blood Transfusion in the Treatment of Cerebral Palsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Xiao Huimei, Professor, Guangdong Women and Children Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GuangdongWCHRD
Record Dates: First submitted 2018-12-18; First posted 2019-01-02 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Safety Issues; Effect of Drugs
Keywords: Cerebral palsy; Autologous Umbilical Cord Blood; safety; effect
MeSH Terms: conditions — Cerebral Palsy | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% sodium chloride infusion any time after entering the Placebo Group, doses is 20-30ml. The infusion speed is 1ml/min.
  Interventions: Drug: 0.9% Sodium Chloride
- Cord Blood Mononuclear Cells(CBMNC) (Experimental): Autologous Umbilical Cord Blood Mononuclear Cells Therapy any time after the diagnosis of cerebral palsy, doses is 20-30ml (total Mononuclear cells>1*10^7/kg). The infusion speed is 1ml/min.
  Interventions: Biological: Autologous Umbilical Cord Blood

INTERVENTIONS:
Drug: 0.9% Sodium Chloride — 0.9% Sodium Chloride in control group
  Arms: Placebo
Biological: Autologous Umbilical Cord Blood — Autologous Umbilical Cord Blood Mononuclear Cells Therapy in Cerebral Palsy for safety and effect evaluation.
  Other Names: Autologous Umbilical Cord Blood Mononuclear Cells Therapy
  Arms: Cord Blood Mononuclear Cells(CBMNC)

SUMMARY:
To study the clinical efficacy and safety of autologous umbilical cord blood transfusion in the treatment of cerebral palsy.

DETAILED DESCRIPTION:
This is a Phase 1 clinical trial that constitutes two time points cohorts with participants who will receive intravenous autologous umbilical cord blood and 0.9% sodium chloride respectively. The timing of treatment is any time after the diagnosis of cerebral palsy. The investigator will proceed the groups during the same period.

1. Demographic Data and Baseline Characteristics of the Studied Group were collected:

   * Basic patient's information survey
   * Medical history
   * Physical examination
   * Basic blood test result
   * Children's developmental disorders evaluation before the treatment
   * Brain Magnetic Resonance Imaging-Diffusion Tensor Imaging (MRI-DTI) before the treatment
   * Neurocognitive function test before the treatment
2. Assessment of clinical condition in the course by measurement of blood pressure, heart and respiratory rates, temperature and adverse events was recorded.
3. Autologous cord blood doses is 20-30ml (total Mononuclear cells>1*10^7/kg)，the infusion speed is 1ml/min, and with same volume of 0.9% sodium chloride as placebo.
4. The follow-up: clinical test until 30th month in 3 month gaps.

ELIGIBILITY:
Inclusion Criteria:

* A patient who was diagnosed with a mild case, and severity case of cerebral palsy or developmental disability through developmental assessment from more than two specialists including a specialist in pediatrics and rehabilitation medicine..
* In case there is a sign of the general decrease in white matter, or periventricular leukomalacia near cerebral ventricles in MRI DTI test.
* A subject who did a written consent to participation in this clinical trial through the very person and a legal representative.

Exclusion Criteria:

* In case a patient underwent a surgical procedure, or was administered autologous cord blood within one year before participating in a clinical trial.
* Accompanied by a serious disease, such as chromosome abnormality, etc.
* In case where a patient's medical condition is judged to be maladapted by a researcher.
* In case a patient or his or her legal representative doesn't agree to participation in a clinical trial.
* A patient having a predisposition to allergies.
* A patient having serious disorders in the liver, kidney, and cardiopulmonary function.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-10-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
The Change of Gross Motor Function Classification System(GMFCS) Score | up to 30 months after therapy at a 3-month interval
  GMFCS is used to assess the gross motor function of the children who were diagnosised as cerebral palsy.The results of GMFCS are divided into five levels. Grade I represents the best outcome while grade Ⅴ represents the worst.
The Change of Gesell Developmental Scale(GDS) Score | every 3-month after therapy until 30 months
  The GDS is used to measure the gross motor,fine action,adaptability，language and individual-society function of the children whose age ranges from 1-month to 6-year-old. The score less than 75 for each subscale represent the worse outcome and more than 75 represent the better.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Yanqun, Phd, Study Director — Guangdong Women and Children Hospital
Locations (1):
- Guangdong Women and Children's Hospital and Health Institute, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun JM, Song AW, Case LE, Mikati MA, Gustafson KE, Simmons R, Goldstein R, Petry J, McLaughlin C, Waters-Pick B, Chen LW, Wease S, Blackwell B, Worley G, Troy J, Kurtzberg J. Effect of Autologous Cord Blood Infusion on Motor Function and Brain Connectivity in Young Children with Cerebral Palsy: A Randomized, Placebo-Controlled Trial. Stem Cells Transl Med. 2017 Dec;6(12):2071-2078. doi: 10.1002/sctm.17-0102. Epub 2017 Oct 28. PMID 29080265